CLINICAL TRIAL: NCT05471908
Title: The Follow-up Automatically vs. As-Needed Comparison Trial
Brief Title: Follow-up Automatically vs. As-Needed Comparison (FAAN-C) Trial
Acronym: FAAN-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Eric Coon, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IHS-2021C1-22388
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia; Urinary Tract Infections; Soft Tissue Infections; Gastroenteritis
Keywords: post-hospitalization; follow-up care; patient centered care; randomized control trial
MeSH Terms: conditions — Pneumonia; Urinary Tract Infections; Soft Tissue Infections; Gastroenteritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Owing to the nature of the comparators, blinding of participants and their medical providers is not possible. However, outcomes that require adjudication will be adjudicated by persons blinded to the subject's randomized group. Outcomes requiring adjudication in FAAN-C are the safety outcomes (hospital readmissions related to the index infection and medical errors). Specifically, a clinician will determine if the readmission was related to the index infection and a separate clinician will score parent-reported medical errors in terms of severity (as described in the Safety Reporting section of the protocol). The clinicians performing adjudication of these outcomes will be blinded to the subject's randomized group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- As-needed (PRN) post-hospitalization follow-up (Experimental): At hospital discharge, participant receives a recommendation for PRN follow-up. Recommendation informs participant that scheduling a follow-up visit is not needed at discharge and suggests that participant follow symptoms after discharge to decide if a visit is ultimately needed or not.
  Interventions: Behavioral: As-needed follow up
- Automatic post-hospitalization follow-up (Active Comparator): At hospital discharge, participant receives a recommendation for automatic follow-up. Recommendation instructs participant to schedule a follow-up visit and attend the visit even if symptoms get better.
  Interventions: Behavioral: Automatic follow-up

INTERVENTIONS:
Behavioral: As-needed follow up — At hospital discharge, participant receives a recommendation for PRN follow-up. Recommendation informs participant that scheduling a follow-up visit is not needed at discharge and suggests that participant follow symptoms after discharge to decide if a visit is ultimately needed or not.
  Other Names: PRN (pro re nata)
  Arms: As-needed (PRN) post-hospitalization follow-up
Behavioral: Automatic follow-up — At hospital discharge, participant receives a recommendation for automatic follow-up. Recommendation instructs participant to schedule a follow-up visit and attend the visit even if symptoms get better.
  Arms: Automatic post-hospitalization follow-up

SUMMARY:
Compare the effectiveness of automatic vs as-needed (PRN) post-hospitalization follow-up for children who are hospitalized for common infections.

DETAILED DESCRIPTION:
BACKGROUND:

Automatic post-hospitalization follow-up visits are commonly recommended by hospital-based pediatricians. The intuitive appeal of automatic follow-up visits is that they might decrease hospital readmissions and promote continuity of care. However, automatic follow-up visits result in missed work for parents, missed school for children, and expenses like co-pays and transportation costs. The principal alternative strategy to automatic follow-up is PRN (pro re nata, "as-needed") follow-up, a patient and family-centered approach that empowers parents to monitor their child's symptoms and decide if a follow-up visit is necessary.

OBJECTIVE:

Compare the effectiveness of automatic vs as-needed (PRN) post-hospitalization follow-up for children who are hospitalized for common infections.

DESIGN:

The Follow-up Automatically vs As-Needed Comparison (FAAN-C, or "fancy") trial is a multicenter randomized controlled trial

POPULATION:

Children hospitalized for pneumonia, skin and soft tissue infection, acute gastroenteritis, or urinary tract infection will be eligible for enrollment.

EXPERIMENTAL INTERVENTION:

Randomization to a recommendation for PRN post-hospitalization follow-up

CONTROL INTERVENTION:

Randomization to a recommendation for automatic post-hospitalization follow-up

OUTCOMES:

The primary outcome is hospital readmission within 14 days of discharge. Secondary outcomes are medical interventions and child health-related quality of life. Exploratory outcomes are cost burden, child time, parent time, symptom duration, total additional ambulatory visits, non-primary care ambulatory visits, parent self-efficacy, parent anxiety, satisfaction with care, telephone and electronic communications with medical providers, well-child visits, immunizations, usual place of medical care, and medical interventions related to the index infection. Safety outcomes are medical errors and hospital readmissions related to the index infection.

TRIAL SIZE:

A total of 2,674 patients (1,337 patients in each group) will be randomized, providing 90% power to demonstrate non-inferiority of a recommendation for PRN follow-up compared to a recommendation for automatic follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years at the time of randomization
* Hospitalization due to a primary diagnosis of pneumonia, skin and soft tissue infection, acute gastroenteritis, or urinary tract infection.
* Parent speaks English or Spanish.

Exclusion Criteria:

* Presence of a comorbid disease that is both chronic and complex
* Principal disease required surgical intervention (beyond superficial incision and drainage)
* Immunodeficiency
* A well-child check-up or post-hospitalization follow-up visit is already scheduled within 7 days of hospital discharge
* Parent or participant strongly prefers PRN or automatic follow-up
* A medical provider feels strongly that a post-hospitalization follow-up visit is needed within 7 days of hospital discharge
* Sibling concurrently hospitalized
* Unable to identify a clinic where the participant would receive any needed post-hospitalization follow-up
* Diagnosis of pneumonia complicated by:

  o Receiving a chest tube
* Diagnosis of urinary tract infection complicated by:

  * History of neurogenic bladder or urologic surgery
  * Renal imaging anticipated within 7 days of hospital discharge
  * Renal abscess
* Diagnosis of skin and soft tissue infection complicated by:

  * Chronic wound
  * Postoperative infection
  * Predisposition to poor wound healing
  * Discharging with a drain in place
  * Complicated by necrotizing fasciitis or toxic shock syndrome
* Diagnosis of gastroenteritis complicated by:

  * Hemolytic uremic syndrome

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2674 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Hospital readmission | Within 14 days of hospital discharge
  The proportion of participants who experience a hospital readmission within 14 days of their index hospital discharge.

SECONDARY OUTCOMES:
Medical interventions | Within 14 days of hospital discharge
  The proportion of participants who receive either a laboratory test, imaging test, or a new medication within 14 days of hospital discharge
Child health-related quality of life | 7 days after hospital discharge
  Mean health-related quality of life score 7 days after hospital discharge, measured by the Impact on Activities and Routines instrument.

OTHER OUTCOMES:
Cost burden | Within 14 days of hospital discharge
  Mean total costs to parents (missed income and expenses) related to the participant's illness within 14 days of hospital discharge, measured by the cost burden survey.
Child time | Within 14 days of hospital discharge
  Mean number of hours of school or daycare missed by the participant within 14 days of hospital discharge as a result of their medical needs
Parent time | Within 14 days of hospital discharge
  Mean number of hours spent away from responsibilities (work or non-work related) by parents within 14 days of hospital discharge as a result of their child's medical needs
Symptom duration | Within 7 days of hospital discharge
  Proportion of participants who have completely recovered from their infection at 7 days after hospital discharge
Total additional ambulatory visits | Within 30 days of hospital discharge
  Mean number of ambulatory visits (in-person or via telehealth) that a participant attends, apart from the post-hospitalization follow-up visit, within 30 days of hospital discharge; Ambulatory visits include clinic, urgent care, and emergency department (not resulting in hospital admission) visits.
Non-primary care ambulatory visits | Within 30 days of hospital discharge
  Mean number of ambulatory visits (in-person or via telehealth) to non-primary care providers, within 30 days of hospital discharge; Non-primary care providers will include all providers outside of the clinic that families identify as their primary care clinic.
Parent self-efficacy | 7 days after hospital discharge
  Mean self-efficacy score 7 days after hospital discharge, measured by the PROMIS self-efficacy short form.
Parent anxiety | 7 days after hospital discharge
  Mean anxiety score 7 days after hospital discharge, measured by the PROMIS anxiety short form.
Satisfaction with care | 7 days after hospital discharge
  Proportion of participants who report agreeing or strongly agreeing with the statement, "I am satisfied with the medical care my child has received since hospital discharge," 7 days after hospital discharge
Telephone and electronic communications with medical providers | Within 14 days of hospital discharge
  Mean number of telephone and electronic (excluding telehealth visits) communications with a medical provider within 14 days of hospital discharge
Well-child visits | Within 6 months of hospital discharge
  Proportion of participants who attend a well-child visit within Proportion of participants who attend a well-child visit within 6 months of hospital discharge
Immunizations | Within 6 months of hospital discharge
  Proportion of participants who receive an immunization within 6 months of hospital discharge
Usual place of medical care | Within 6 months of hospital discharge
  Proportion of participants who report having a usual place of medical care 6 months after hospital discharge
Medical interventions related to the index infection | Within 14 days of hospital discharge
  Proportion of participants who receive either a laboratory test, imaging test, or a new medication related to the index infection within 14 days of hospital discharge
Medical errors | Within 14 days of hospital discharge
  Proportion of parents who report that their child experienced a medical error within 14 days of hospital discharge, measured by the Family Safety Interview
Hospital readmissions related to the index infection | Within 14 days of hospital discharge
  Proportion of participants who experience a hospital readmission related to the index infection within 14 days of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eric Coon, MD, Principal Investigator — University of Utah
Locations (14):
- United States (14):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Packard at El Camino Hospital, Mountain View, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - St. Louis Children's Hospital, St Louis, Missouri
  - Penn Medicine Princeton Medical Center, Plainsboro, New Jersey
  - Cincinnati Children's Hospital Medical Center - Main Campus, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center - Liberty Campus, Liberty Township, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Main, Houston, Texas
  - Texas Children's West, Houston, Texas
  - Intermountain Primary Children's Hospital Larry H. and Gail Miller Family Campus, Lehi, Utah
  - Riverton Hospital, Riverton, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT05471908/Prot_001.pdf